CLINICAL TRIAL: NCT03274232
Title: Efficacy and Tolerance of an Injectable Medical Device Containing Hyaluronic Acid and Amino Acids: a Monocentric Six-month Open-label Evaluation
Brief Title: Face Photoaging: Efficacy and Tolerance Evaluation of an Intradermal Injective Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DERMING E0916
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-07

CONDITIONS: Face Skin Photoaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SUNEKOS ® 200 (Experimental): The 1st intradermal treatment (T1i) was performed during the basal visit (T0), after basal evaluations planned by the study procedure and repeated after 10 (T2i), 20 (T3i) and 30 (T4i) days.
  Interventions: Device: SUNEKOS ® 200

INTERVENTIONS:
Device: SUNEKOS ® 200 — micro-injections of the study product were performed by a specialized dermatologist, bilaterally on the face (zygomatic protuberance, nostril's angle, inferior margin of tragus, lip marionette lines, mandibular angle) of female volunteers aged 45-65 years, with photoaging of mild/moderate grade

SUMMARY:
Efficacy and tolerance evaluation of an intradermal injective treatment

DETAILED DESCRIPTION:
Primary end point of the study was to evaluate clinically and by non-invasive instrumental evaluations tolerance and efficacy of SUNEKOS ® 200 injectable treatment on main sign of face skin photoaging; the micro-injections of the study product were performed by a specialized dermatologist, bilaterally on the face (zygomatic protuberance, nostril's angle, inferior margin of tragus, lip marionette lines, mandibular angle) of female volunteers aged 45-65 years, with photoaging of mild/moderate grade.

ELIGIBILITY:
Inclusion Criteria:

* - female sex;
* age 45-65 years;
* mild/moderate cutaneous photoaging according to a reference photographic scale (see Appendix 8)
* skin phototype I, II and III according to Fitzpatrick's classification, with a preference to grade II-III (see par. 8.1)
* agreeing to present at each study visit without make-up;
* accepting to not change their habits regarding food, physical activity, make-up use, face cosmetic and cleansing products;
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes), during the entire duration of the study;
* accepting to sign the Informed consent form.

Exclusion Criteria:

* Dependent on the volunteers' characteristics
* Pregnancy;
* lactation;
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* Body Mass Index (BMI) variation (± 1) during the study period;
* subjects not in menopause who do not accept to perform the pregnancy test during the basal visit, 30 days (T4i) and 2 months (T2M) after the first biomineralizing treatment execution;
* performing skin treatments for aesthetic correction (biomaterials implants, face lifting, botox injections, laser, chemical peeling) in the 12 months prior to the study start;
* performing permanent filler in the past;
* change in the normal habits regarding food, physical activity, face cosmetic, cleansing and make-up use during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study actually or during the previous 6 months.
* Presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.).
* Diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* pulmonary disease
* cancer
* neurological or psychological disease
* inflammatory/immunosuppressive disease
* drug allergy.
* Anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* assumption of drugs able to influence the test results in the investigator opinion.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Variation of Wrinkle Severity Rating Scale (WSRS) grade | Basal visit (T0), 10 days(T2i), 20 days (T3i), 30 days (T4i), 2 months (T2M) , 3 months (T3M), 6 months (T6M)
  Reduction of wrinkles severity corresponding to a decrease from the baseline of the Wrinkle Severity Rating Scale (WSRS) clinical score where:
  Grade 1 (absent): no visible nasolabial fold; continuous skin line. Grade 2 (mild): shallow but visible nasolabial fold with a slight indentation; minor facial feature.
  Grade 3 (moderate): moderately deep nasolabial folds; clear facial feature visible at normal appearance but not when stretched.
  Grade 4 (severe): very long and deep nasolabial folds; prominent facial feature; <2mm visible fold when stretched.
  Grade 5 (very severe): extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched.
Variation of Facial Volume Loss Scale (FVLS) grade | Basal visit (T0), 10 days(T2i), 20 days (T3i), 30 days (T4i), 2 months (T2M) , 3 months (T3M), 6 months (T6M)
  Reduction of face volume loss corresponding to a decrease from the baseline of the Facial Volume Loss Scale (FVLS) where Grade 1 Mild flattening or shadowing of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). No prominent bony landmarks. No visibility of underlying musculature.
  Grade 2 An intermediate point between grade 1 and grade 3. Grade 3 Moderate concavity of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas. Prominence of bony landmarks. May have visibility of underlying musculature.
  Grade 4 An intermediate point between grade 3 and grade 5. Grade 5 Severe indentation of one or more facial regions (including the cheek, temple, preauricolar and periorbital areas). Severe prominence of bony landmarks. Clear visibility of underlying musculature.

SECONDARY OUTCOMES:
Superficial skin hydration variation | Basal visit (T0), 2 months (T2M) , 3 months (T3M), 6 months (T6M)
  Improvement of skin electrical capacitance value measured with Corneometer CM825 (Courage - Khazaka, Köln, Germany).
  The measure of the skin capacitance properties is an indirect expression of its hydration level.
Deep skin hydration variation | Basal visit (T0), 2 months (T2M) , 3 months (T3M), 6 months (T6M)
  Improvement of tissue dielectric constant value of superficial and deep skin layers measured with MoistureMeterD (Delfin Technologies, Kuopio - Finland)
Skin plastoelasticity variation | Basal visit (T0), 2 months (T2M) , 3 months (T3M), 6 months (T6M)
  Improvement of the principal torsiometric parameters Ue (immediate extensibility), Uf (final extensibility), Uv (viscoelasticity) and Ur (immediate elastic recovery).Skin firmness is measured with the instrument Dermal Torque Meter (Dia-Stron Ltd., UK).
Variation of profilometric parameters | Basal visit (T0), 2 months (T2M) , 3 months (T3M), 6 months (T6M)
  Reduction of the crow's feet lines profilometric parameters versus baseline where Ra is average roughness of the analysed profile, Rt is wrinkles total high, Rv is wrinkles maximum depth.
Photographic documentation (3D pictures ) | Basal visit (T0), 2 months (T2M) , 3 months (T3M), 6 months (T6M)
  Three-dimensional pictures of the face taken by VECTRA H1 handheld imaging system.
Face volume variation | Basal visit (T0), 2 months (T2M) , 3 months (T3M), 6 months (T6M)
  Face volume image analysis was carried on the 3D pictures taken by Vectra H1 thanks to Vectra analysis module (VAM) software